CLINICAL TRIAL: NCT01157559
Title: Efficacy and Safety With Ziprasidone in the Treatment of First-episode Schizophrenia Spectrum Disorder: Multi-center Study
Brief Title: Efficacy and Safety With Ziprasidone in First-episode Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Young Chul Chung/Professor of Psychiatry, Chonbuk National University Hospital, Jeonju, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-Zeldox in FEP
Record Dates: First submitted 2010-06-30; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2007-01

CONDITIONS: First Episode Psychosis
MeSH Terms: interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ziprasidone — 8 week prospective study

SUMMARY:
The aim of the study is to investigate the efficacy and safety of ziprasidone in patients with first episode psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet DSM-IV criteria for first episode schizophrenia, schizophreniform disorder and schizoaffective disorder

Exclusion Criteria:

* Patients with previously prescribed antipsychotic medication in 2 weeks or more
* patients with substance-induced psychotic disorder, serious suicide attempt, neurological disorder, etc.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Primary Completion 2008-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Symptoms assessment by objective rating scales | week 1
  PANSS total score, SANS, clinical global impression scale, GAF
Symptoms assessment by objective rating scales | week 2
  PANSS total score, SANS, clinical global impression scale, GAF
Symptoms assessment by objective rating scales | week 4
  PANSS total score, SANS, clinical global impression scale, GAF
Symptoms assessment by objective rating scales | week 6
  PANSS total score, SANS, clinical global impression scale, GAF
Symptoms assessment by objective rating scales | week 8
  PANSS total score, SANS, clinical global impression scale, GAF, DAS-S

SECONDARY OUTCOMES:
Assessment of adverse events by objective rating scales and self report scales | one-month
  Simpson and Angus rating scale, Barnes Akathisia rating scale and Abnormal Involuntary Movement Scale
Assessment of adverse events by objective rating scales and self report scales | two-month.
  Simpson and Angus rating scale, Barnes Akathisia rating scale and Abnormal Involuntary Movement Scale

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Department of Psychiatry, Chonbuk national University Hospital, Jeonju
  - Heo psychiatric Hospital, Jeonju
  - Jeonju Jesus Hospital, Jeonju